CLINICAL TRIAL: NCT05337228
Title: A Randomized, Open-label, Multi-center Phase III Clinical Trial to Evaluate the Safety and Efficacy of IN-C006 Peri Inj. Compared With RPN301 in Postoperative Patients Requiring Peripheral Parenteral Nutrition
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of IN-C006 Peri Inj. Compared With RPN301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IN_PPN_301
Record Dates: First submitted 2022-03-28; First posted 2022-04-20 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-02

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IN-C006 Peri inj. (Experimental): IN-C006 Peri inj. 1904 mL
  Interventions: Drug: IN-C006 Peri inj.
- RPN301 (Active Comparator): RPN301 2020 mL
  Interventions: Drug: RPN301

INTERVENTIONS:
Drug: IN-C006 Peri inj. — IN-C006 peri inj. will be injected continuously for 3 days.
  Arms: IN-C006 Peri inj.
Drug: RPN301 — RPN301 will be injected continuously for 3 days.
  Arms: RPN301

SUMMARY:
This study is designed to evaluate the safety and efficacy of IN-C006 Peri inj. and RPN301 in postoperative patients requiring central parenteral nutrition.

DETAILED DESCRIPTION:
This study is a randomized, open-label, phase 3 design. The subject will be assigned to one of the two treatment groups (IN-C006 Peri inj. or RPN301)

ELIGIBILITY:
Inclusion Criteria:

* Age over 19 at the time of obtaining the informed consent form
* Requiring over 3 days of parenteral nutrition via a peripheral vein after an operation
* BMI 16 ~ 30 kg/㎡

Exclusion Criteria:

* Has received parenteral nutrition within 7 days of screening
* Severe dyslipidemia
* Uncontrolled diabetes
* Clinically significant liver disease
* Clinically significant kidney disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Adverse drug reaction rate | Day 1 to Day 4
  Rate of treatment-related adverse events as assessed by CTCAE v5.0 and investigator's evaluation

SECONDARY OUTCOMES:
Change in nutritional management parameters(Nitrogen balance) | Day 1 to Day 4
  Nitrogen balance(Nitrogen intake-Nitrogen out)
Change in nutritional management parameters(Prealbumin) | Day 1 to Day 4
  Prealbumin(mg/L)
Change in nutritional management parameters(Albumin) | Day 1 to Day 4
  Albumin(g/dL)
Change in nutritional management parameters(Transferrin) | Day 1 to Day 4
  Transferrin(mg/dL)
Change in inflammation parameters(hs-CRP) | Day 1 to Day 4
  hs-CRP(mg/L)
Change in inflammation parameters(TNF-α) | Day 1 to Day 4
  TNF-α(pg/mL)
Change in inflammation parameters(IL-6) | Day 1 to Day 4
  IL-6(pg/mL)
Change in fatty acid profile | Day 1 to Day 4
  LA(ug/mL), AA(ug/mL), EPA(ug/mL), DHA(ug/mL)
Incidence of Adverse event | Day 1 to Day 4
  Rate of adverse events as assessed by CTCAE v5.0 and investigator's evaluation
Change in laboratory parameters (Hematology) | Day 1 to Day 4
  Difference in the proportion of subjects whose test results changed from normal to abnormal between the IN-C006 Peri group and the RPN301 group
  - Hematology
Change in laboratory parameters (Blood chemistry) | Day 1 to Day 4
  Difference in the proportion of subjects whose test results changed from normal to abnormal between the IN-C006 Peri group and the RPN301 group
  - Blood chemistry
Change in laboratory parameters (Blood coagulation test) | Day 1 to Day 4
  Difference in the proportion of subjects whose test results changed from normal to abnormal between the IN-C006 Peri group and the RPN301 group
  - Blood coagulation test
Change in laboratory parameters (Urinalysis) | Day 1 to Day 4
  Difference in the proportion of subjects whose test results changed from normal to abnormal between the IN-C006 Peri group and the RPN301 group
  - Urinalysis
Change in vital sign (Blood pressure) | Day 1 to Day 4
  Changes between the IN-C006 Peri group and the RPN301 group (mean difference at the last visit compared to the Baseline (Day 1))
  - Systolic blood pressure(mmHg), Diastolic blood pressure(mmHg)
Change in vital sign (Pulse rate) | Day 1 to Day 4
  Changes between the IN-C006 Peri group and the RPN301 group (mean difference at the last visit compared to the Baseline (Day 1))
  - Pulse rate(rate)
Change in vital sign (Body temperature) | Day 1 to Day 4
  Changes between the IN-C006 Peri group and the RPN301 group (mean difference at the last visit compared to the Baseline (Day 1))
  - Body temperature(℃)
Change in vital sign (Respiratory rate) | Day 1 to Day 4
  Changes between the IN-C006 Peri group and the RPN301 group (mean difference at the last visit compared to the Baseline (Day 1))
  - Respiratory rate(rate)
Normal and abnormal change in physical examination (Frequency) | Day 1 to Day 4
  Frequency of subjects who were normal/clinically insignificant abnormalities before administration of investigational products to clinically significant abnormalities at least once after administration of investigational products
  - General Appearance, HEENT (Head, Eyes, Ears, Nose, Throat), Skin (including hair, nails), Respiratory, Cardiovascular, Chest/Lungs/Breast, Abdominal/Gastrointestinal, Musculoskeletal, Extremities/Joint, Neurological/Psychological, Lymph nodes, Rectal/Pelvic/Genitalia, Other
Normal and abnormal change in physical examination (Ratio) | Day 1 to Day 4
  Ratio of subjects who were normal/clinically insignificant abnormalities before administration of investigational products to clinically significant abnormalities at least once after administration of investigational products
  - General Appearance, HEENT (Head, Eyes, Ears, Nose, Throat), Skin (including hair, nails), Respiratory, Cardiovascular, Chest/Lungs/Breast, Abdominal/Gastrointestinal, Musculoskeletal, Extremities/Joint, Neurological/Psychological, Lymph nodes, Rectal/Pelvic/Genitalia, Other

CONTACTS AND LOCATIONS:
Overall Officials: Do Joong PARK, Study Chair — Seoul National Univerity Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No